CLINICAL TRIAL: NCT06499532
Title: The Frequency of Trigeminocardiac Reflex During the Extraction of Impacted Mandibular Wisdom Teeth and the Effect of Anesthesia Technique on the Development of the Reflex
Brief Title: The Frequency of Trigeminocardiac Reflex During the Extraction of Impacted Mandibular Wisdom Teeth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kutahya Health Sciences University (Other)
Responsible Party: Principal Investigator, Bedreddin Cavlı, Assistant Professor Doctor, Kutahya Health Sciences University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Screening
Other Study IDs: KutahyaHSU/BedreddinCavli/001
Record Dates: First submitted 2024-06-30; First posted 2024-07-12 (Actual); Last update posted 2024-07-12 (Actual); Status verified 2024-07

CONDITIONS: Trigemino-Cardiac Reflex; Impacted Third Molar Tooth
Keywords: Trigemino-Cardiac Reflex,; Impacted Third Molar Tooth; Hemodynamic instability

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Gow-gates anesthesia, distance to inferior alveolar nerve is more than 1 mm (Experimental): The extraction of impacted wisdom teeth in patients forming this study arm was performed using the Gow-Gates anesthesia technique. In these patients, the distance between the wisdom teeth and the inferior alveolar nerve is greater than 1 mm.
  Interventions: Procedure: Monitoring and Surgical removal of mandibular impacted wisdom teeth, using Gow-Gates anesthesia technique
- Gow-gates anesthesia, distance to inferior alveolar nerve is less than 1 mm (Experimental): The extraction of impacted wisdom teeth in patients forming this study arm was performed using the Gow-Gates anesthesia technique. In these patients, the distance between the wisdom teeth and the inferior alveolar nerve is less than 1 mm.
  Interventions: Procedure: Monitoring and Surgical removal of mandibular impacted wisdom teeth, using Gow-Gates anesthesia technique
- İnferior alveoler nerve block,distance to inferior alveolar nerve is more than 1 mm (Experimental): The extraction of impacted wisdom teeth in patients forming this study arm was performed using the inferior alveolar nerve block technique and supplemental anesthesia (buccal- mylohyoid). In these patients, the distance between the wisdom teeth and the inferior alveolar nerve is greater than 1 mm.
  Interventions: Procedure: Monitoring and Surgical removal of mandibular impacted wisdom teeth, using inferior alveolar nerve block anesthesia technique
- İnferior alveoler nerve block, distance to inferior alveolar nerve is less than 1 mm (Experimental): The extraction of impacted wisdom teeth in patients forming this study arm was performed using the inferior alveolar nerve block technique and supplemental anesthesia (buccal- mylohyoid). In these patients, the distance between the wisdom teeth and the inferior alveolar nerve is less than 1 mm.
  Interventions: Procedure: Monitoring and Surgical removal of mandibular impacted wisdom teeth, using inferior alveolar nerve block anesthesia technique

INTERVENTIONS:
Procedure: Monitoring and Surgical removal of mandibular impacted wisdom teeth, using Gow-Gates anesthesia technique — The surgical removal of impacted mandibular wisdom teeth in patients included in the study arms was performed using Gow-Gates anesthesia technique. Patients were monitored for TCR during the procedure.
  Arms: Gow-gates anesthesia, distance to inferior alveolar nerve is less than 1 mm; Gow-gates anesthesia, distance to inferior alveolar nerve is more than 1 mm
Procedure: Monitoring and Surgical removal of mandibular impacted wisdom teeth, using inferior alveolar nerve block anesthesia technique — The surgical removal of impacted mandibular wisdom teeth in patients included in the study arms was performed using inferior alveolar nerve block anesthesia technique and supplemental anesthesia (buccal- mylohyoid). Patients were monitored for TCR during the procedure.
  Arms: İnferior alveoler nerve block, distance to inferior alveolar nerve is less than 1 mm; İnferior alveoler nerve block,distance to inferior alveolar nerve is more than 1 mm

SUMMARY:
The goal of this clinical trial is to investigate trigeminocardiac reflex (TCR) formation during surgical extraction of mandibular impacted wisdom teeth in healthy adults. The main questions it aims to answer are:

* How often is the TCR encountered during the extraction of impacted mandibular wisdom teeth?
* Do different local anesthesia techniques affect the frequency of this reflex?
* Is the relationship between the impacted teeth and the inferior alveolar nerve a predisposing factor for the development of this reflex

Researchers will monitor patients included in the study during the extraction of impacted mandibular wisdom teeth.

Patients will undergo an anxiety test, and those found to be anxious will be excluded from the study (to avoid vasovagal events).

During the procedure, at seven different surgical stages, blood pressure, oxygen saturation, and heart rate data will be recorded at the beginning and end of each stage.

The monitoring of TCR was conducted by observing a sudden bradycardia that developed within a few seconds and resolved when the procedure was paused, not preceded by any tachycardia. TCR will be investigated at three different levels according to different reference values in the literature.

DETAILED DESCRIPTION:
The study included 40 patients who underwent extraction of impacted mandibular wisdom teeth.Before the surgical procedure, the two most commonly used local anesthesia techniques in oral surgical practice, GG and IASB techniques, were applied. While IASB was always accompanied by buccal and mylohyoid area supportive anesthesia, no additional anesthesia was required in any patient receiving GG anesthesia. Evaluation of the patients was done using panoramic radiographs. The closest distance between the roots of the relevant wisdom teeth and the inferior alveolar nerve (IAN) was recorded. In cases where the distance was less than 1 mm or where superimposition occurred, cone beam computed tomography (CBCT) images were taken from the patients to confirm the distance in three dimensions.

Patients were divided into two groups based on the proximity of their wisdom tooth roots to the IAN (within 1 mm or more than 1 mm) and into two groups based on the anesthesia technique to be applied (GG-IASB). Subgroups were named as GG-0 (more than 1 mm from IAN), GG-1 (within 1 mm from IAN), IASB-0 (more than 1 mm from IAN), and IASB-1 (within 1 mm from IAN). Ten patients were evenly selected for each subgroup (GG-0, GG-1, IASB-0, IASB-1).

The surgeries included in the study were performed by a single surgeon. Impacted wisdom teeth were vertical and consisted of teeth retained in bone. For the surgical procedure, a sleeve flap was applied including distal horizontal and vertical relaxing incisions near the mesial papilla of mandibular second molar tooth.

TCR monitoring was conducted by observing the occurrence of sudden bradycardia, which could develop within a few seconds and show improvement upon pausing the procedure, not preceded by tachycardia. To ensure accurate and timely monitoring of this sudden process and to monitor potential asystole that could develop, patients were monitored. Monitoring was conducted using 5-channel Contec Medical Systems (Hebei, China) monitors. Throughout the procedure, heart rate, systolic blood pressure (SBP), diastolic blood pressure (DBP), mean arterial pressure, and oxygen saturation were recorded. Records were taken at six separate surgical stages: initially during local anesthesia administration, and subsequently during incision/flap removal, removal of bone barriers, crown elevation, root elevation, and during suturing. Any sudden changes occurring during the procedure were recorded along with their onset times.

In defining TCR (Trigeminocardiac Reflex) in the literature, various reference measurement methods include sudden drops in heart rate by more than 10%, more than 20%, or dropping below 60 beats per minute. To highlight these different proportional reference drop values, severity grading was used in the observed TCR findings. Sudden drops in heart rate between 10% and 20% were classified as mild TCR (TKR-1), drops exceeding 20% and heart rate falling below 60 bpm as moderate TCR (TKR-2), and the presence of asystole, syncope, or need for atropine application as severe TCR (TKR-3). The total TCR across all grades was termed as t-TCR. TCR calculation was based on heart rate measurements taken at the beginning of each surgical stage.

To exclude vasovagal syncope, commonly cited as a neurological emergency and etiological factor, and high anxiety from the study, patients were initially subjected to anxiety tests, and individuals with high anxiety levels were excluded from the study. Patient anxiety levels were assessed using the Amsterdam Preoperative Anxiety and Information Scale (APAIS) and the State-Trait Anxiety Inventory-State scale (STAI-S).

ELIGIBILITY:
Inclusion Criteria:

* 18-30 years old
* Will have impacted tooth extraction for the first time
* Extraction indication for mandibular impacted wisdom teeth
* Systemically healthy individuals

Exclusion Criteria:

* Patients with high anxiety
* Female patients who are pregnant or breastfeeding
* Individuals with any systemic disease
* Individuals with suspicion of cysts and/or tumors in the area of mandibular impacted wisdom teeth
* Patients with mental or neurological disorders
* Patients using antidepressants

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2023-10-01 (Actual); Primary Completion 2023-11-01 (Actual); Study Completion 2023-11-10 (Actual)

PRIMARY OUTCOMES:
Heart rate monitoring | During the operation
  All patients in all research arms monitored prior to extraction of impacted mandibular wisdom teeth had their heart rate monitored throughout the procedure.
Systolic, and diastolic blood pressure monitoring | During the operation
  All patients in all research arms monitored prior to extraction of impacted mandibular wisdom teeth had their systolic, and diastolic blood pressure monitored throughout the procedure.
Oxygen saturation monitoring | During the operation
  All patients in all research arms monitored prior to extraction of impacted mandibular wisdom teeth had their oxygen saturation monitored throughout the procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Bedreddin Cavlı, Asst. Professor, Principal Investigator — Kutahya University of Health Sciences
Locations (1):
- Kutahya University of Health Sciences, Kütahya, Turkey (Türkiye)

DOCUMENTS (1):
  • Study Protocol (2023-10-01): https://cdn.clinicaltrials.gov/large-docs/32/NCT06499532/Prot_000.pdf